CLINICAL TRIAL: NCT05855304
Title: Comparison Of The Sacroiliac Manipulation And Kinesiological Tape In Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: basketball tape and manupila
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: balance; jump
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual therapy (Experimental)
  Interventions: Other: manual therapy
- Kinesiology taping (Experimental)
  Interventions: Other: Kinesiology taping

INTERVENTIONS:
Other: manual therapy — The leg length was measured while the subjects were lying on their stomachs. Then, by grasping the lateral malleolus, the knees are bent 90 degrees and changes in leg length were observed, the positions of the SI joints were noted. Afterwards, the person
  Arms: manual therapy
Other: Kinesiology taping — As part of the tape (kinesio tex brand) kinesio protocol used in this study, the starting position of the kinesio tape is the site of lumbar spine flexion. Kinesio tape was applied transversely to the bilateral sacroiliac joint area as a long I-shaped piece of tape with 80% tension and no tension was applied to the ends of the tape. Another short tape will be adhered to the SI joint with 80% tension at a right angle to the hip, and no tension is applied to the ends of the tape.
  Arms: Kinesiology taping

SUMMARY:
In the USA, basketball is the most popular team sport for boys and girls enrolled in the 2003-2004 school year. Many countries offer opportunities for young people to learn the game in a variety of settings, from physical education classes, school competitions, public and private sports organizations to community entertainment programmes. While the USA has long been seen as the dominant power in basketball, recent results in competitions such as the 1988 and 2004 Men's Olympic Games and 2002 World Championships show the rest of the world is closing the gap. Basketball continues to spread around the world, thanks to ongoing development programs for children and youth .

DETAILED DESCRIPTION:
One of the important parameters of postural control during landing after jump is stabilization time. There are several studies proving the curative effect of kinesio taping. However, studies investigating the effect of sacroiliac chiropractic manipulation are more limited than kinesio taping studies. There are fewer studies evaluating the performance of trait juvenile basketball players. Although there is evidence showing the effect of manipulation on performance, Botelho et al. state that scientific evidence in this area is lacking.

ELIGIBILITY:
Inclusion criteria

* Being a licensed basketball player in amateur leagues in Istanbul
* Being between the ages of 18-25
* Being a man
* Voluntarily participating in the study
* Not having a verbal communication barrier

Exclusion criteria

* Being under 18 years old or over 25 years old
* Spondylolysis or spondylolisthesis
* Neurological problems (acute myelopathy, spinal cord compression, cauda equina syndrome, radicular impingement)
* Hypermobile joints
* Acute fractures
* Intracanalicular hematomas
* Spinal cord hematomas in the spine
* Postoperative fixation prostheses
* Neoplastic diseases of muscle or other tissues
* To have a surgical operation on the knee and waist region in the last year
* Osteoporosis with risk of fracture
* Vertebrobasilar insufficiency

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Jump | one day
  The optojump system will be used in this study as a jumping power measurement tool.
  In the measurements, the vertical jump height was recorded with the optoJump system and the software of this system (Microgate, Bolzano, Italy). The measurement of the vertical jump distance in centimeters is done by means of two bars in the OptoJump system with sensors that detect movement. The duration of the jump (milliseconds) is also included in determining the jump distance.
patrick faber test | one day
  The person to be tested is in the supine position, while the practitioner is standing next to the patient. The practitioner applies some pressure over the bent knee towards the bed. The force applied in this position is thought to exert pressure on the anterior SI ligaments and hip joint.
Derifield leg check | one day
  If the leg, which is observed to be short in the prone position, is observed to be extended compared to the previous state when the knees are extended 90 degrees, the test is called positive derifield.
  When the applied person is in the prone position and the knees are brought to the 90 degree flexion position, the short observed leg is again observed to be short or if it is found to be even shorter, it is called a negative derifield.

SECONDARY OUTCOMES:
Yeoman's test | one day
  The tester supports the SI joint with one hand and grasps the knee on the same side with the other, and lifts the hip off the bed. Since tension will occur in the anterior sacroiliac ligament in this position, pain in the SI joint indicates a positive test.
Gillet test | one month
  The Gillet test is used to evaluate the mobility of the SI joint. While the person to be treated is standing, the practitioner is behind the person to be tested. The practitioner places one finger on the SIPS and the other finger on the 2nd sacral processus spinosus. The SIPS is expected to move down while the patient raises one knee.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Torres-Ronda L, Ric A, Llabres-Torres I, de Las Heras B, Schelling I Del Alcazar X. Position-Dependent Cardiovascular Response and Time-Motion Analysis During Training Drills and Friendly Matches in Elite Male Basketball Players. J Strength Cond Res. 2016 Jan;30(1):60-70. doi: 10.1519/JSC.0000000000001043. PMID 26284807